CLINICAL TRIAL: NCT02224716
Title: Multicenter Intervention Program to Optimize the Clinical Management of Community-acquired Pneumonia in Hospitals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Other Study IDs: FIS-ANT-2014-01
Record Dates: First submitted 2014-08-22; First posted 2014-08-25 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Community Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-intervention All patients admitted with a diagnosis of CAP
- Post intervention All patient admitted with a diagnosis of CAP

SUMMARY:
The purpose of this study is to evaluate the impact of a structured package (bundle) in reducing the use of antimicrobials and hospital stay of patients with community-acquired pneumonia (CAP), and no increase in mortality of these patients in different hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CAP at hospital admission .
* Age: 18 years or more.

Exclusion Criteria:

* Patients with nosocomial pneumonia or criteria related to health care.
* Patients with severe immunosuppression (HIV infection with <200 CD4+ lymphocytes / mm3), neutropenia (<500 neutrophils / mm3).
* Patient treated with immunosuppressive drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre-intervention period
  All patients admitted with a diagnosis of CAP will be included in the participating centers during the 12 months prior to the intervention. Case detection is done through the electronic record of the basic minimum data set (MDS) (2, 36). Diagnosed patients will be selected at discharge: "simple acute bronchitis and pneumonia excluding asthma major criteria" (by diagnosis related group, DRG 541) and "simple and pleuritis in over 17 Pneumonia" (DRG 089).
  Post-intervention period
  All patients admitted with a diagnosis of CAP in the participating centers, which measures the bundle will apply prospectively included. Case detection was performed by daily review of patients admitted to target units and will be coordinated by the IP address of each center.
Sampling Method: Non-Probability Sample
Enrollment: 968 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Antimicrobial use in patients hospitalized for CAP. | twelve months
  It is measured in defined daily doses (DDD) per 100 hospital stay of patients hospitalized with CAP.
Mortality rate to 30 days | twelve months
  Number of death of patients hospitalized with CAP, stratified by CURB-65 score.

SECONDARY OUTCOMES:
CAP severity CURB-65 or PSI registered. | twelve months
  Implementation of quality indicators in the management of CAP. They are expressed as dichotomous variables (yes / no):
  Numbers of doctors who register on the clinical history the evaluation of CAP severity by CURB-65 or PSI at hospitalization.
Microbiological samples at admission. | twelve months
  Implementation of quality indicators in the management of CAP. They are expressed as dichotomous variables (yes / no):
  Numbers of doctors who taking all microbiological samples recommended in the guideline in the first 6 hours of patient admission.
Appropriate supportive treatment | Twelve months
  Implementation of quality indicators in the management of CAP. They are expressed as dichotomous variables (yes / no):
  Number of doctors who take supportive treatment according to guideline during the hospitalization.
Empirical treatment | Twelve months
  Implementation of quality indicators in the management of CAP. They are expressed as dichotomous variables (yes / no):
  Number of doctors who prescribed empirical treatment according to the guideline at admission.
Appropriate sequential therapy. | Twelve months
  Implementation of quality indicators in the management of CAP. They are expressed as dichotomous variables (yes / no):
  Number of doctors who switch to oral therapy according to guideline.
Specific antimicrobial treatment | Twelve months
  Implementation of quality indicators in the management of CAP. They are expressed as dichotomous variables (yes / no):
  Number of doctors who prescribed the specific antimicrobial treatment defined in the guideline
Total duration of antibiotic therapy. | Twelve months
  Implementation of quality indicators in the management of CAP. They are expressed as dichotomous variables (yes / no):
  Number of doctors who prescribe an antimicrobial treatment during 7 days or less, or 5 days or less after clinical improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Retamar Gentil, Study Director — Hospital Universitario Virgen Macarena; Juan Enrique Corzo Delgado, Principal Investigator — Hospital Universitario Virgen de Valme; Cristina Roca Oporto, Principal Investigator — Hospitales Universitarios Virgen del Rocío; Montserrat Pérez Pérez, Principal Investigator — Hospital de la Línea de la Concepción; Salvador López Cardenas, Principal Investigator — Hospital de Jerez de la Frontera; María del Carmen Almodóvar Pulido, Principal Investigator — Hospital de Antequera; Fernando Nebrera Navarro, Principal Investigator — Hospital de Formentera; Rosario Javier Martínez, Principal Investigator — University Hospital Virgen de las Nieves; Francisca Guerrero Sánchez, Principal Investigator — Hospital Universitario Puerta del Mar
Locations (1):
- Fundación Pública Progreso y Salud, Seville, Sevilla, Spain